CLINICAL TRIAL: NCT00237887
Title: A Phase III, Multicenter Study of the Efficacy and Safety of Adalimumab Treatment in Subjects With Moderate to Severe Chronic Plaque Psoriasis
Brief Title: Efficacy and Safety of Adalimumab in Subjects With Moderate to Severe Chronic Plaque Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M03-656
Record Dates: First submitted 2005-10-07; First posted 2005-10-13 (Estimated); Last update posted 2007-08-29 (Estimated); Status verified 2007-08

CONDITIONS: Psoriasis
Keywords: Psoriasis; adalimumab
MeSH Terms: conditions — Psoriasis | interventions — Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: adalimumab

SUMMARY:
A Phase III, Multicenter Study of the Efficacy and Safety of Adalimumab Treatment in Subjects with Moderate to Severe Chronic Plaque Psoriasis

ELIGIBILITY:
Inclusion Criteria:

* Subject was age 18 or older and in good health (Investigator discretion) with a recent stable medical history.
* Subject had a clinical diagnosis of psoriasis for at least 6 months, had moderate to severe plaque psoriasis.
* Subject was able and willing to self-administer sc injections or had available qualified person(s) to administer sc injections

Exclusion Criteria:

* Subject had previously received anti-TNF therapy.
* Subject cannot discontinue systemic therapies and/or topical therapies for the treatment of psoriasis and cannot avoid UVB or PUVA phototherapy
* Subject cannot avoid excessive sun exposure
* Subject is taking or requires oral or injectable corticosteroids
* Subject considered by the investigator, for any reason, to be an unsuitable candidate for the study
* Female subject who is pregnant or breast-feeding or considering becoming pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1212 (Actual)
Dates: Start 2004-12

PRIMARY OUTCOMES:
Proportion of subjects achieving clinical response at Week 16 relative to the Baseline (Week 0) PASI score | Week 16

SECONDARY OUTCOMES:
Safety parameters

CONTACTS AND LOCATIONS:
Overall Officials: Beverly Paperiello, Study Director — Abbott

REFERENCES:
- [Derived] Armstrong AW, Villanueva Quintero DG, Echeverria CM, Gu Y, Karunaratne M, Reyes Servin O. Body Region Involvement and Quality of Life in Psoriasis: Analysis of a Randomized Controlled Trial of Adalimumab. Am J Clin Dermatol. 2016 Dec;17(6):691-699. doi: 10.1007/s40257-016-0229-x. PMID 27815915
- [Derived] Papp KA, Armstrong AW, Reich K, Karunaratne M, Valdecantos W. Adalimumab Efficacy in Patients with Psoriasis Who Received or Did Not Respond to Prior Systemic Therapy: A Pooled Post Hoc Analysis of Results from Three Double-Blind, Placebo-Controlled Clinical Trials. Am J Clin Dermatol. 2016 Feb;17(1):79-86. doi: 10.1007/s40257-015-0161-5. PMID 26547918
- [Derived] Gordon K, Papp K, Poulin Y, Gu Y, Rozzo S, Sasso EH. Long-term efficacy and safety of adalimumab in patients with moderate to severe psoriasis treated continuously over 3 years: results from an open-label extension study for patients from REVEAL. J Am Acad Dermatol. 2012 Feb;66(2):241-51. doi: 10.1016/j.jaad.2010.12.005. Epub 2011 Jul 14. PMID 21752491
- [Derived] Revicki DA, Menter A, Feldman S, Kimel M, Harnam N, Willian MK. Adalimumab improves health-related quality of life in patients with moderate to severe plaque psoriasis compared with the United States general population norms: results from a randomized, controlled Phase III study. Health Qual Life Outcomes. 2008 Oct 2;6:75. doi: 10.1186/1477-7525-6-75. PMID 18831744
- [Derived] Menter A, Tyring SK, Gordon K, Kimball AB, Leonardi CL, Langley RG, Strober BE, Kaul M, Gu Y, Okun M, Papp K. Adalimumab therapy for moderate to severe psoriasis: A randomized, controlled phase III trial. J Am Acad Dermatol. 2008 Jan;58(1):106-15. doi: 10.1016/j.jaad.2007.09.010. Epub 2007 Oct 23. PMID 17936411